CLINICAL TRIAL: NCT02174120
Title: The Application of Target Controlled Infusion of Etomidate Combined With Propofol in the Maintenance of Anesthesia During Brain Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu He, Physician, Henan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140623
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Target Controlled Infusion; General Anesthesia
MeSH Terms: interventions — Propofol; Etomidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): During maintenance of anesthesia, etomidate was give by target controlled infusion, the effect-site concentration is 0.3 to 0.6 micrograms/ml to keep bispectral index between 40 to 60.
  Interventions: Drug: etomidate
- Group B (Experimental): During maintenance of anesthesia, Propofol was give by target controlled infusion, the effect-site concentration is 2 to 4 micrograms/ml to keep bispectral index between 40 to 60.
  Interventions: Drug: propofol
- Group C (Experimental): During maintenance of anesthesia, etomidate will be given by target controlled infusion for 2 h first, and then propofol will be given by target controlled infusion, the effect-site concentration is 0.3 to 0.6 micrograms/ml and 2 to 4 micrograms/ml, respectively. Bispectral index should be kept between 40 to 60.
  Interventions: Drug: propofol; Drug: etomidate

INTERVENTIONS:
Drug: propofol
  Arms: Group B; Group C
Drug: etomidate
  Other Names: Fu Er Li
  Arms: Group A; Group C

SUMMARY:
To explore the application of target controlled infusion of etomidate combined with propofol in the maintenance of anesthesia during brain surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60 and 80 years Brain surgeries Body weight is between 45 to 75 kg and body mass index is no more than 30 kg/m2 American Society of Anesthesiology (ASA) Physical Status: Ⅰ or Ⅱ Expected operation duration is between 3 and 5 h Signed informed consent form

Exclusion Criteria:

* Serious cardiac, cerebral(acute stroke, uncontrolled seizure, sever dementia), liver, kidney, lung, endocrine disease or sepsis History of general anesthesia within 24 h before the operation Long use of hormone or history of adrenal suppression Hyperlipidaemia Long use of psychotropic substances Systolic pressure is still under 90 mm Hg after twice given of vasopressor agent Suspected abuse of narcotic analgesia Patients need to use neuromuscular blocking drugs (except intubation) Allergy to trial drug or other contraindication Pregnant or breast-feeding women Attendance of other trial past 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Baseline to the end of the operation, expected to be about 6 h
  Heart rate should be recorded before induction, 1 min, 5 min, 20 min after intubation, at the time of skin incision, skull drilling, incision of dura matter, during intracranial operation, suture of dura matter and skin.
Blood pressure | Baseline to the end of the operation, expected to be about 6 h
  Blood pressure should be recorded before induction, 1 min, 5 min, 20 min after intubation, at the time of skin incision, skull drilling, incision of dura matter, during intracranial operation, suture of dura matter and skin.
Concentration of cortisol | from baseline to the end of the operation, expected to be about 6 h
  Concentration of cortisol should be recorded before induction, 30 min, 1 h, 2 h after intubation, and immediately when the operation is over.

SECONDARY OUTCOMES:
Use of vasoactive agent | from the beginning of induction to the end of the operation, expected to be about 6 h
  The name and dose of the vasoactive agents used from the beginning of induction to the end of operation.
The time from stop of remifentanil to awake | The time from stop of remifentanil to awake, expected to no more than 15 min
Severity of agitation | Within 24 h after the operation
Postoperative nausea and vomiting | Within 24 h after the operation
Dose of etomidate and propofol | From the beginning of induction to the end of the operation, expected to be about 6 h
Intraoperative awareness | From the beginning of induction to the end of the operation, expected to be about 6 h
Expense of anesthetics | From the beginning of induction to the end of the operation, expected to be about 6 h
Allergic reaction | From beginning of induction to 24 h after the operation